CLINICAL TRIAL: NCT00400283
Title: A Randomised, Double-blind, Placebo-controlled, Multiple Oral Dose, Dose Escalation Trial, Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC 55-0414 in Patients With Type 2 Diabetes
Brief Title: A Study Looking Into the Effect of NNC 55-0414 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN414-1384
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NNC 55-0414

SUMMARY:
This trial is conducted in Europe. A seven day dose escalation study in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diet treatment only for at least two weeks
* Body mass index (BMI) between 22-34 kg/m2 inclusive
* HbA1C between 6.5-12.0% inclusive
* Fasting blood glucose (FBG) between 7.0-18.0 mmol/L inclusive
* Patients should be negative (lesser than 70 kU/l) for antibodies against glutamic acid decarboxylase (GAD)

Exclusion Criteria:

* Pharmacological treatment with medication or pancreatitis that the Investigator expected to interfere with blood glucose levels
* History of cancer or any clinically significant cardiovascular respiratory, hepatic, haematological, gastrointestinal, dermatological, venereal, neurological or psychiatric disorder as judged by the Investigator
* Impaired renal function, serum creatinine greater than 150µmol/L
* Patients, who were known to have serum hepatitis or who were carriers of the Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies, or had a positive result to the test for HIV 1/2 antibodies
* Patients, who had received an investigational drug in the four months new chemical entity or licensed product preceding the start of dosing
* Patients, who had donated plasma or blood in the past month, or in excess of 500 mL in the past 12 weeks
* Patients who had a significant history of alcoholism or drug/chemical abuse

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-01-19 (Actual); Primary Completion 2001-05-03 (Actual); Study Completion 2001-05-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety and the tolerability of ascending multiple oral doses of NNC 55 0414 in patients with type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com